CLINICAL TRIAL: NCT02715791
Title: Teams Advancing Patient Experience: Strengthening Quality for People Through Health Connectors for Diabetes Management (TAPESTRY-HC-DM): A Feasibility RCT
Brief Title: TAPESTRY With Health Connnectors for Diabetes Management
Acronym: TAP-HC-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Health Canada (Other Government); McMaster Family Health Team (Unknown); Volunteer Hamilton (Unknown); INSPIRE-PHC (Unknown)
Responsible Party: Principal Investigator, Gina Agarwal, Associate Professor, Department of Family Medicine, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0744
Record Dates: First submitted 2015-11-03; First posted 2016-03-22 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes Mellitus; Hypertension
Keywords: Self-Management; Health Connectors; Volunteers; Technology; Interprofessional team; Chronic disease; Self-efficacy; Patient-centredness; Community Engagement
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Other): Patients randomized to the control group will receive usual care and upon the end of study will receive access to the Healthy Lifestyle App and the McMaster PHR
  Interventions: Other: Usual Care
- TAP-HC-DM (Other): Patients randomized to the intervention group will get TAP-HC-DM intervention from time zero
  Interventions: Behavioral: TAP-HC-DM

INTERVENTIONS:
Behavioral: TAP-HC-DM — Patients randomized to the intervention group will complete the Healthy Lifestyle App modules. Their results will create a report with a suggested list of tip sheets that patients, volunteers, and clinics will see.
  Patients will also be encouraged to access the McMaster PHR in order to track their health, and communicate with volunteers or the clinic.
  Volunteer health connectors will connect with patients at least weekly, by phone, McMaster PHR message, or in person (depending on patient preference). They will be motivating, providing tip sheets or other education, doing tech support, providing community resources, and building a volunteer-patient relationship with the client.
  Clinicians will see and triage the reports, and may follow up on various aspects identified.
  Arms: TAP-HC-DM
Other: Usual Care — Patients randomized to the control group will receive usual care and upon the end of the intervention arm of the study will receive the TAPESTRY-HC-DM intervention as detailed in the intervention group.
  Arms: Usual Care

SUMMARY:
The TAPESTRY-HC-DM approach is designed to support self-management of chronic disease by strengthening connections between patients and the primary healthcare system through "health connectors" -both volunteers and technology including the TAPESTRY Healthy Lifestyle App and McMaster Personal Health Record (PHR). It will explore whether strengthening primary care connections across patients, providers, and community organizations through TAPESTRY-HC-DM - i.e., the deployment of volunteer health connectors coordinated by a community organization, the use of the TAPESTRY Healthy Lifestyle e-Application by patients, and care coordination processes by the interprofessional primary healthcare team - can increase self-efficacy in managing chronic conditions.

DETAILED DESCRIPTION:
TAP-HC-DM is a feasibility randomized controlled trial (RCT) involving various pieces of intervention and their interactions to form a complex adaptive system. The purpose of the trial is to assess the effectiveness of the intervention not only through evaluating patient outcomes, but also through understanding the process of implementation and its fidelity to core elements.

The trial will be conducted within the McMaster Family Health Team (MFHT) in Hamilton, Ontario. The MFHT consists of two sites, with approximately 30,000 patients, as well as 30 family physicians, 70 family medicine residents, 10 nurse practitioners and other healthcare professionals.

Initial lists of potential participants will be created using an algorithm based on the inclusion criteria that will be run on the clinics' electronic medical records systems, with manual chart audits completed afterwards on an as-needed basis. The family physicians will then be asked to vet this list for further exclusion criteria. Patients from the list will then be sent a package including an invite letter from their family physician and a consent form.

Participants who have consented, will receive a welcome call from volunteers who will then provide detailed description of the program and expectations. The clients will then be invited to sign up for McMaster Personal Health Record (PHR) and asked to complete the modules (Diabetes, Hypertension, Sleep, Exercise, Nutrition, Medications, PHR) on the Healthy Lifestyle app. After completion of the modules, participants will receive a report and suggested tip sheets based on their responses. Volunteers as health connectors will connect with clients weekly, providing motivation, education, tech support, and community connections. The healthcare teams at the clinics will also receive the report and will triage it in their weekly huddles. Any follow-up recommended by the clinics will be communicated to volunteers who will then work with clients on the given recommendations, or directly to patients.

ELIGIBILITY:
Inclusion Criteria:

* Active patient at McMaster Family Health Team
* Aged 18+
* Diagnosis of Diabetes
* Diagnosis of Hypertension
* Regular access to a computer

And at least ONE of:

* Uncontrolled HbA1C measures (in the past 6 months, or most recent) - 10
* Uncontrolled recent blood pressure (in the past 3 months, or most recent) - 140/90 or higher (either number higher)
* Newly diagnosed with diabetes (diagnosed within 6 months)
* End-stage organ damage/other complications of diabetes [e.g. renal dysfunction, diabetic neuropathy]
* Doctor Recommendation

Exclusion Criteria:

* identified as deceased
* explicitly stated they do not want to be part of a research project
* reside in long-term care
* are receiving end-of-life care
* directly related to anyone from the McMaster University Department of Family Medicine
* not a participant in another TAPESTRY project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2017-09-26 (Actual)

PRIMARY OUTCOMES:
Diabetes self-efficacy | 4-month
  This is the primary outcome which will be measured by Stanford Diabetes Self-Efficacy Scale, an 8-item scale.

SECONDARY OUTCOMES:
Self-efficacy in Managing General Chronic Conditions | 4-month
  The outcome will be measured by a 6-item Stanford Self-Efficacy Scale for Managing Chronic Disease. It covers several domains that are common across many chronic diseases, symptom control, role function, emotional functioning and communicating with physicians.
Attainment of Health Goals | 4-month
  The outcome will be assessed using a Goal Attainment Scale (GAS) Questionnaire
Assessment of Care for Chronic Conditions | 4-month
  The outcome will be assessed using Assessment of Care for Chronic Conditions survey having 20 items
Patient Empowerment | 4-month
  The outcome will be assessed using Patient Empowerment questionnaire, a 5-item survey questionnaire and Canadian Institutes of Health Research (CIHR) Common Indicator for the Community- Based Primary Health Care (CBPHC)
Patient Centredness | 4-month
  The outcome will be assessed using Patient Centeredness questionnaire, a 6-item questionnaire and CIHR Common Indicator for the Community- Based Primary Health Care (CBPHC)
Satisfaction with Healthcare | 4-month
  This will be measured using a one item questionnaire that inquires how clients would like to rate the quality of healthcare they received on a scale of 0-100 (0=not satisfied, 100=completely satisfied)
Patient Activation | 4-month
  This will be assessed by a 13-item Patient Activation Measure (PAM) questionnaire.
Patient Readiness for Change | 4-month
  Readiness-for-Change Questionnaire (RCQ) for Diabetes Self-Management will be used to examine the clients' stage of readiness for diabetes management behaviour change (pre-contemplation, contemplation, action, maintenance), developed based on the Cardiovascular Risk Reduction Program Readiness-to-Change Lifestyle Behavior
Physical Activity | 4-month
  This will be assessed using the Rapid Assessment of Physical Activity (RAPA).

CONTACTS AND LOCATIONS:
Overall Officials: David Price, MD, CCFP, Study Chair — Professor and Chair, McMaster Department of Family Medicine; Lisa Dolovich, PharmD, MSc, Principal Investigator — Co-Principal Investigator, McMaster Department of Family Medicine
Locations (3):
- Canada (3):
  - McMaster Family Health Practice, Hamilton, Ontario
  - McMaster University Department of Family Medicine, Hamilton, Ontario
  - Stonechurch Family Health Centre, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agarwal G, Gaber J, Richardson J, Mangin D, Ploeg J, Valaitis R, Reid GJ, Lamarche L, Parascandalo F, Javadi D, O'Reilly D, Dolovich L. Pilot randomized controlled trial of a complex intervention for diabetes self-management supported by volunteers, technology, and interprofessional primary health care teams. Pilot Feasibility Stud. 2019 Oct 27;5:118. doi: 10.1186/s40814-019-0504-8. eCollection 2019. PMID 31673398